CLINICAL TRIAL: NCT06933407
Title: This Study Investigates the Role of Strain Elastography in Assessing Paraurethral Tissue Elasticity in Continent and Incontinent Pre- and Postmenopausal Women. It Also Evaluates the Predictive Value of Strain Elastography Compared to Other Pelvic Imaging Modalities, Including Conventional Ultrasound Examinations, in Supporting Treatment Decision-making for Urinary Incontinence.
Brief Title: Elastographic Assessment of Suburethral Tissue in Continent and Incontinent Women
Acronym: SE-inc1
Status: Recruiting | Type: Observational
Sponsor: Szeged University (Other)
Collaborators: Capio Specialized Center for Gynecology, Solna, 182 88 Stockholm, Sweden (Unknown)
Responsible Party: Principal Investigator, Dr. Csákány Lóránt, Head of the Urogynecology Outpatient Clinic, Szeged University
Other Study IDs: 55/2016
Record Dates: First submitted 2025-03-20; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence (UI); Urinary Bladder, Overactive; Incontinence, Overactive Bladder, Stress Urinary Incontinence; Stress Urinary Incontinence (SUI)
Keywords: Urinary Incontinence; Bladder dysfunction; Urine leakage; Stress urinary incontinence (SUI)
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Control group (asymptomatic women): This group consists of women without any symptoms of urinary incontinence. They serve as a baseline for comparison with the affected groups. No specific intervention is applied to this group.
  Interventions: Diagnostic Test: Strain Elastography
- Stress urinary incontinence (SUI) group: This group includes women diagnosed with stress urinary incontinence (SUI), characterized by involuntary urine leakage during physical exertion, coughing, sneezing, or other activities that increase intra-abdominal pressure.
  Interventions: Diagnostic Test: Strain Elastography
- Stress urinary incontinence (SUI) with hypermobile urethra: This subgroup includes women with stress urinary incontinence and hypermobility of the urethra, which is assessed through clinical examination and/or imaging techniques.
  Interventions: Diagnostic Test: Strain Elastography
- Stress urinary incontinence (SUI) without hypermobile urethra: This subgroup consists of women with stress urinary incontinence but without significant urethral hypermobility. The absence of hypermobility may suggest intrinsic sphincter deficiency (ISD) as a primary factor in incontinence.
  Interventions: Diagnostic Test: Strain Elastography
- Stress urinary incontinence (SUI) group without estrogen therapy: Women diagnosed with stress urinary incontinence (SUI) who do not receive vaginal estrogen therapy. This group will serve as a reference to assess the natural biomechanical properties of paraurethral tissues in SUI patients.
  Interventions: Diagnostic Test: Strain Elastography
- Stress urinary incontinence (SUI) group with estrogen therapy: Women diagnosed with stress urinary incontinence (SUI) who undergo vaginal estrogen therapy as part of their treatment. This group will be evaluated to determine the effects of vaginal estrogen on paraurethral tissue elasticity and its potential role in improving urethral support and biomechanical properties.
  Interventions: Diagnostic Test: Strain Elastography

INTERVENTIONS:
Diagnostic Test: Strain Elastography — Strain elastography (SE) is a parametric imaging modality that assesses tissue deformation in response to externally applied pressure, providing qualitative and semi-quantitative information on tissue elasticity and mechanical properties. Unlike conventional 2D ultrasound, SE enables the objective evaluation of paraurethral tissue stiffness, which may play a role in the pathophysiology of stress urinary incontinence (SUI). SE will be performed on three predefined paraurethral regions to assess pelvic floor elasticity and biomechanical characteristics. A standardized protocol will be implemented to ensure high reproducibility, with controlled probe compression and precisely defined regions of interest. SE may improve the diagnostic accuracy and therapeutic decision-making for SUI by identifying differences in tissue compliance among affected women.

SUMMARY:
Strain elastography (SE) will be utilized as a non-invasive imaging technique to evaluate tissue elasticity and biomechanical properties in women with stress urinary incontinence (SUI) and in continent controls. The primary aim is to determine whether SE can detect differences in paraurethral tissue stiffness between these groups. Given the established role of tissue elasticity in the pathophysiology of SUI, SE will be investigated as a potential diagnostic tool in urogynecological evaluations.

This prospective cohort study will be conducted at a tertiary referral center. All participants will undergo introital two-dimensional (2D) ultrasound in the midsagittal plane at rest. SE will be performed in three predefined suburethral regions of interest (ROIs):

* internal urethral orifice (IUO) level
* midurethra (MU) level
* external urethral orifice (EUO) level

The adipose layer (AL) between the external urethral meatus and the pubic symphysis will serve as the reference tissue, representing the softest anatomical structure in the region.

Descriptive and comparative statistical analyses will be conducted to assess differences in paraurethral tissue stiffness between the study groups.

It is hypothesized that SE will be able to detect differences in paraurethral tissue elasticity, with SUI being associated with increased tissue compliance. The study also aims to determine whether SE can reliably distinguish between varying degrees of tissue stiffness in women with SUI and continent controls.

Pathophysiological focus:

The study will explore key mechanisms underlying SUI, including:

* Weakened bladder neck support
* Impaired urethral stabilization due to increased tissue elasticity and collagen degradation
* While conventional 2D ultrasound provides anatomical information, it does not directly evaluate tissue biomechanics. In contrast, SE enables real-time visualization of tissue elasticity, offering a promising adjunct to traditional urogynecological assessment methods.

Standardization and Protocol

The study will follow a standardized protocol to ensure reproducibility and high-quality data. Key methodological elements include:

* Minimal probe compression during introital ultrasound to avoid artifacts
* Bladder emptying prior to examination to eliminate confounding effects
* Carefully standardized ROI placement across all patients
* Controlled image acquisition conditions to reduce variability

Future Directions

* Future research based on this study will aim to:
* Optimize SE protocols and refine ROI placement strategies
* Establish clinical cutoff values for differentiating tissue stiffness in SUI vs. continent women
* Assess the long-term effects of pelvic floor muscle training (PFMT) and vaginal estrogen therapy on paraurethral biomechanics
* Facilitate the integration of SE into routine urogynecological practice to support early diagnosis and personalized treatment strategies for SUI

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stress urinary incontinence (SUI) based on patient history, physical examination, and/or urodynamic assessment.

Exclusion Criteria:

* Pelvic malignancy or history of pelvic radiation therapy
* Urge urinary incontinence (UUI) or detrusor overactivity
* Pelvic organ prolapse (POP) stage ≥ II (based on POP-Q classification)
* Pregnancy or recent postpartum status (less than 6 months postpartum)
* Neurological disorders affecting bladder function
* Recurrent urinary tract infections (UTIs) or active lower urinary tract infection
* Inability to undergo study procedures
* Cognitive impairment or psychiatric conditions affecting informed consent or compliance

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will include adult women in Hungary diagnosed with stress urinary incontinence (SUI), along with a control group of continent women. Participants will be recruited from urogynecology outpatient clinics, tertiary referral centers, and gynecology departments.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Paraurethral Tissue Elasticity in Women with Stress Urinary Incontinence Using Strain Elastography | At a single study visit, within two weeks of enrollment.
  Detection of a statistically significant difference in paraurethral tissue elasticity between women with stress urinary incontinence (SUI) and continent controls using strain elastography (SE), with high measurement reproducibility across predefined regions of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- University of szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Quantitative strain elastography measurements of periurethral tissue elasticity.

REFERENCES:
- [Background] Falconer C, Ekman-Ordeberg G, Ulmsten U, Westergren-Thorsson G, Barchan K, Malmstrom A. Changes in paraurethral connective tissue at menopause are counteracted by estrogen. Maturitas. 1996 Jul;24(3):197-204. doi: 10.1016/s0378-5122(96)82010-x. PMID 8844634
- [Background] Tunn R, Petri E. Introital and transvaginal ultrasound as the main tool in the assessment of urogenital and pelvic floor dysfunction: an imaging panel and practical approach. Ultrasound Obstet Gynecol. 2003 Aug;22(2):205-13. doi: 10.1002/uog.189. PMID 12905521
- [Background] DeLancey JO. Structural support of the urethra as it relates to stress urinary incontinence: the hammock hypothesis. Am J Obstet Gynecol. 1994 Jun;170(6):1713-20; discussion 1720-3. doi: 10.1016/s0002-9378(94)70346-9. PMID 8203431
- [Background] Kreutzkamp JM, Schafer SD, Amler S, Strube F, Kiesel L, Schmitz R. Strain Elastography as a New Method for Assessing Pelvic Floor Biomechanics. Ultrasound Med Biol. 2017 Apr;43(4):868-872. doi: 10.1016/j.ultrasmedbio.2016.12.004. Epub 2017 Jan 17. PMID 28108041
- [Background] Zhao B, Wen L, Chen W, Qing Z, Liu D, Liu M. A Preliminary Study on Quantitative Quality Measurements of the Urethral Rhabdosphincter Muscle by Supersonic Shear Wave Imaging in Women With Stress Urinary Incontinence. J Ultrasound Med. 2020 Aug;39(8):1615-1621. doi: 10.1002/jum.15255. Epub 2020 Mar 3. PMID 32125001
- [Background] Falah-Hassani K, Reeves J, Shiri R, Hickling D, McLean L. The pathophysiology of stress urinary incontinence: a systematic review and meta-analysis. Int Urogynecol J. 2021 Mar;32(3):501-552. doi: 10.1007/s00192-020-04622-9. Epub 2021 Jan 8. PMID 33416968
- [Background] Patel UJ, Godecker AL, Giles DL, Brown HW. Updated Prevalence of Urinary Incontinence in Women: 2015-2018 National Population-Based Survey Data. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):181-187. doi: 10.1097/SPV.0000000000001127. Epub 2022 Jan 12. PMID 35030139